CLINICAL TRIAL: NCT03220256
Title: Protocol Establishment for the Prevention of Lamotrigine-induced Skin Rash in Epilepsy Patients: A Pilot Study
Brief Title: Protocol Establishment for the Prevention of Lamotrigine-induced Skin Rash in Epilepsy Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Kun Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1605-121-764
Record Dates: First submitted 2017-07-12; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Lamotrigine Allergy
MeSH Terms: interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lamotrigine tolerance (Experimental): The dose of lamotrigine (0.1mg) started to increase and gradually increased according to the drug tolerance induction protocol, and the efficacy was evaluated by dosing to the commercial capacity (100mg bid) within 2 weeks.
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — The dose of lamotrigine (0.1mg) started to increase and gradually increased according to the drug tolerance induction protocol, and the efficacy was evaluated by dosing to the commercial capacity (100mg bid) within 2 weeks. In addition, the ratio of regulatory T cells was measured before lamotrigine administration, and the proportion of regulatory T cells was measured by two-week administration of lamotrigine after tolerance induction protocol. Add 6 ml of EDTA tube to each cryovial, and dispense 1 ml each in cryovial. After the appropriate number of patients of the same phenotype were collected, the analysis was performed.

SUMMARY:
The investigators intend to find a way to lower drug rash occurrence by applying drug tolerance induction protocol at the beginning of lamotrigine administration.

Genotyping of participants with rash and those without rash after taking lamotrigine and genetic testing to find common gene mutations in these participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-85 years old
* Epilepsy patients
* Patients who started Lamotrigine first time

Exclusion Criteria:

* Those who do not agree with prior consent
* Women taking oral contraceptives.
* history of drug rash
* Taking enzyme-inducing antiepileptic drugs (EIAED) or valproate (VPA)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08-02 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Skin rash incidence rate | 2 weeks

SECONDARY OUTCOMES:
Changes in Treg cell ratio in peripheral blood | 2 weeks
Severity of skin rash (CTCAE version 4.0) | 2 weeks
Lamotrigine drug level in blood (mcg/ml) | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Wang XQ, Xiong J, Xu WH, Yu SY, Huang XS, Zhang JT, Tian CL, Huang DH, Jia WQ, Lang SY. Risk of a lamotrigine-related skin rash: current meta-analysis and postmarketing cohort analysis. Seizure. 2015 Feb;25:52-61. doi: 10.1016/j.seizure.2014.12.001. Epub 2014 Dec 23. PMID 25645637
- [Background] Murray TS, Rice TW, Wheeler AP, Phillips EJ, Dworski RT, Stollings JL. Medication Desensitization: Characterization of Outcomes and Risk Factors for Reactions. Ann Pharmacother. 2016 Mar;50(3):203-8. doi: 10.1177/1060028015625660. Epub 2016 Jan 18. PMID 26783356
- [Background] Castells M. Desensitization for drug allergy. Curr Opin Allergy Clin Immunol. 2006 Dec;6(6):476-81. doi: 10.1097/ACI.0b013e3280108716. PMID 17088655
- [Background] Akdis CA. Therapies for allergic inflammation: refining strategies to induce tolerance. Nat Med. 2012 May 4;18(5):736-49. doi: 10.1038/nm.2754. PMID 22561837